CLINICAL TRIAL: NCT00002557
Title: PROTOCOL FOR THE MANAGEMENT OF MYCOSIS FUNGOIDES AND THE SEZARY SYNDROME
Brief Title: Combination Chemotherapy in Patients With Advanced or Recurrent Mycosis Fungoides
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000063440; SAFR-CT-MF-2; NCI-F94-0015
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2000-08

CONDITIONS: Lymphoma
Keywords: stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Cutaneous | interventions — VAP-cyclo protocol; Doxorubicin; Etoposide; Leucovorin; Methotrexate

INTERVENTIONS:
Drug: CHOP regimen
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: leucovorin calcium
Drug: methotrexate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of etoposide with or without doxorubicin and methotrexate in treating patients who have mycosis fungoides.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the response rate in patients with Stage III/IV or recurrent mycosis fungoides or Sezary syndrome treated with oral etoposide, with the addition of doxorubicin, then methotrexate for poor responders. II. Assess changes in the hematologic and immunologic status of the tumor in these patients.

OUTLINE: Patients are treated sequentially on Regimens A, B, and C depending on response. The following acronyms are used: CF Leucovorin calcium, NSC-3590 DOX Doxorubicin, NSC-123127 MTX Methotrexate, NSC-740 VP-16 Etoposide, NSC-141540 Regimen A: Single-Agent Chemotherapy. VP-16. Regimen B: 2-Drug Combination Chemotherapy. VP-16/DOX. Regimen C: 3-Drug Combination Chemotherapy. VP-16/DOX/MTX.

PROJECTED ACCRUAL: Study duration will be at least 3 years with an anticipated accrual of 3 patients/year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Stage III/IV mycosis fungoides or Sezary syndrome Stage I/II cutaneous T-cell lymphoma in relapse following interferon therapy also eligible

PATIENT CHARACTERISTICS: Age: Not specified

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior interferon alpha for Stage I/II disease allowed Chemotherapy: Prior isotretinoin for Stage I/II disease allowed Endocrine therapy: Prior topical steroids for Stage I/II disease allowed Radiotherapy: Prior ultraviolet therapy for Stage I/II disease allowed Prior x-ray therapy for Stage I/II disease allowed Surgery: Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 1993-06

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Novitzky, MD, PhD, Study Chair — University of Cape Town
Locations (1):
- University of Cape Town School of Medicine, Cape Town, South Africa